CLINICAL TRIAL: NCT04652661
Title: Intranasal Dexmedetomidine Versus Intranasal Midazolam as Sole Sedative Agents for MRI In Pediatrics: A Randomized Double-Blind Trial
Brief Title: Intranasal Dexmedetomidine Versus Intranasal Midazolam for MRI In Pediatrics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Taysser Mahmoud Abdalraheem, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 32466/11/20
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Dexmedetomidine; Midazolam; MRI; Pediatrics
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Intervention Model Description: Sixty children will be randomly allocated into two equal groups by computer generated sequence through sealed opaque envelopes:
  Group D: 30 children will be sedated with 2 μg/kg intranasal DEX. Group M: 30 children will be sedated with 0.3 mg/kg intranasal midazolam.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Group (Experimental): 30 children will be sedated with 2 μg/kg intranasal dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- Midazolam Group (Active Comparator): 30 children will be sedated with 0.3 mg/kg intranasal midazolam.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — 30 children will be sedated with 2 μg/kg intranasal DEX.
  Arms: Dexmedetomidine Group
Drug: Midazolam — 30 children will be sedated with 0.3 mg/kg intranasal midazolam.
  Arms: Midazolam Group

SUMMARY:
An increasing number of studies have reported the use of dexmedetomidine in clinical practice. However, few studies have reported on the intranasal use of dexmedetomidine in radiological procedures The aim of this work is to compare the efficacy and safety of intranasal dexmedetomidine and intranasal midazolam in pediatrics undergoing MRI.

DETAILED DESCRIPTION:
This prospective randomized double-blind clinical trial will be carried out on 60 children undergoing elective MRI in Tanta University Hospitals.

Sixty children will be randomly allocated into two equal groups by computer-generated sequence through sealed opaque envelopes:

Group D: 30 children will be sedated with 2 μg/kg intranasal DEX. Group M: 30 children will be sedated with 0.3 mg/kg intranasal midazolam.

ELIGIBILITY:
Inclusion Criteria:

Aged from 2 to 8 years Both sexes ASA physical status I and II Elective MRI.

Exclusion Criteria:

1. Patient's guardian refusal.
2. Body mass index >30 kg/m2
3. Known allergy to dexmedetomidine or midazolam.
4. Suspected difficult airway.
5. Upper respiratory tract infection
6. Anatomical structural deformity of the nasal cavity.
7. Severe liver or renal impairment.
8. Severe bradycardia or atrioventricular block above II degree type 2.
9. Administration of digoxin or beta blockers

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
The incidence of successful sedation | One hour
  Successful sedation is defined as the time taken to achieve an MOAA/S score of 4 and is the time when the patients are calm and sedated and allow intravenous cannulation and MRI examination without crying or agitation.

SECONDARY OUTCOMES:
The onset time of sedation | One hour
  The onset time of sedation is defined as the time from drug administration to successful sedation.
The occurrence of Adverse effects | One hour
  The occurrences of adverse events will be recorded (e.g. bradycardia, a significant oxygen saturation decrease, severe arrhythmia or arrest).
The degree of operator satisfaction | One hour
  MRI operator satisfaction before discharge using a 5- point score, with (0 = very dissatisfied, 1 = dissatisfied, 2 = neither satisfied nor dissatisfied, 3 = satisfied and 4 = very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: No
The data will be provided with a reasonable request from authors